CLINICAL TRIAL: NCT06479564
Title: Effects of Free Weight and Machine Training With and Without Aerobic Training on Strength, Endurance and Muscle Mass of Lower Limb Among Body Builders.
Brief Title: Effects of Free Weight and Machine Training With and Without Aerobic Training Among Body Builders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0472
Record Dates: First submitted 2024-06-24; First posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Sports Physical Therapy
Keywords: Resistance Training; Free weights; Machine training; Body Builders
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: randomized control design
Who Masked: Participant
Masking Description: the participants are blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): 20 participants will be in control group, they will only perform free weight training and machine training and will not perform aerobic exercises
  Interventions: Other: free weight training and machine training
- Group B (Experimental): 20 participants will be in experimental group, they will perform aerobic exercises along with free weight training and machine training
  Interventions: Other: Aerobic Exercises

INTERVENTIONS:
Other: free weight training and machine training — 20 participants will be in control group who will only perform free weight and machine training
  Arms: Group A
Other: Aerobic Exercises — 20 participants will be in experimental group giving them aerobic exercise training protocol along with free weight and machine training
  Arms: Group B

SUMMARY:
Effects of free weight and machine training with and without aerobic training among body builders.

DETAILED DESCRIPTION:
Effects of free weight and machine training with and without aerobic training on strength, endurance and muscle mass of lower limb among body builders.

ELIGIBILITY:
Inclusion Criteria:

* Age: - 17-35 years(16)
* Body builders(16)
* Physically fit Athletes (17)
* Male athletes
* Benchmarks for body builders

  1. Minimum 60 kg leg press
  2. Minimum 15 kg hams curl
  3. Minimum 10 kg weighted squats

Exclusion Criteria:

* Participants who will be unable to complete the training
* No musculoskeletal disorder
* No cardiorespiratory disorder
* Jumper's knee
* Any respiratory issue
* Foot and ankle injuries
* Patellar tendinopathy
* Pulmonary disorder
* Ligamentous and meniscal injury
* Bone deformity
* Fractures of lower limb

Ages: 17 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2023-11-23 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
1 Repetition Maximum | 8 weeks
  A 1 Repetition Maximum (1 RM) test is a commonly used method in the fitness and strength training realm to assess an individual's maximum strength for a specific exercise. (18) The test involves determining the maximum amount of weight a person can lift for a single repetition of a given exercise.
Yo-Yo test | 8 weeks
  The 20-meter multistage shuttle test, also known as the "Beep Test" or "Yo-Yo Test," is a commonly used aerobic fitness test. (20)The test involves continuous running between two lines 20 meters apart in response to audio signals. . If a participant fails to reach the line before the beep, they are given a warning. After a second warning, the test is concluded, and the level reached is recorded.
Muscle Mass | 8 weeks
  Measuring muscle size using an inches tape, also known as a tailor's tape or a body tape measure, is a simple and effective way to track changes in muscle size and monitor your fitness progress

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Ibtisam, DPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Sports Academy, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schott N, Johnen B, Holfelder B. Effects of free weights and machine training on muscular strength in high-functioning older adults. Exp Gerontol. 2019 Jul 15;122:15-24. doi: 10.1016/j.exger.2019.03.012. Epub 2019 Apr 10. PMID 30980922
- [Background] Schwanbeck SR, Cornish SM, Barss T, Chilibeck PD. Effects of Training With Free Weights Versus Machines on Muscle Mass, Strength, Free Testosterone, and Free Cortisol Levels. J Strength Cond Res. 2020 Jul;34(7):1851-1859. doi: 10.1519/JSC.0000000000003349. PMID 32358310
- [Background] Alves RC, Prestes J, Enes A, de Moraes WMA, Trindade TB, de Salles BF, Aragon AA, Souza-Junior TP. Training Programs Designed for Muscle Hypertrophy in Bodybuilders: A Narrative Review. Sports (Basel). 2020 Nov 18;8(11):149. doi: 10.3390/sports8110149. PMID 33218168
- [Background] Hackett DA, Johnson NA, Chow CM. Training practices and ergogenic aids used by male bodybuilders. J Strength Cond Res. 2013 Jun;27(6):1609-17. doi: 10.1519/JSC.0b013e318271272a. PMID 22990567
- [Background] Zangene AR, Abbasi A, Nazarpour K. Estimation of Lower Limb Kinematics during Squat Task in Different Loading Using sEMG Activity and Deep Recurrent Neural Networks. Sensors (Basel). 2021 Nov 23;21(23):7773. doi: 10.3390/s21237773. PMID 34883777
- [Background] Imbach F, Sutton-Charani N, Montmain J, Candau R, Perrey S. The Use of Fitness-Fatigue Models for Sport Performance Modelling: Conceptual Issues and Contributions from Machine-Learning. Sports Med Open. 2022 Mar 3;8(1):29. doi: 10.1186/s40798-022-00426-x. PMID 35239054
- [Background] Sun M, Wang L. Effect of Bodybuilding and Fitness Exercise on Physical Fitness Based on Deep Learning. Emerg Med Int. 2022 Jun 21;2022:3891109. doi: 10.1155/2022/3891109. eCollection 2022. PMID 35774151
- [Background] Condello G, Minganti C, Lupo C, Benvenuti C, Pacini D, Tessitore A. Evaluation of change-of-direction movements in young rugby players. Int J Sports Physiol Perform. 2013 Jan;8(1):52-6. doi: 10.1123/ijspp.8.1.52. Epub 2012 Jul 31. PMID 22869638